CLINICAL TRIAL: NCT02069353
Title: Augmented Multimodal Neurologic Monitoring in High Risk Survivors of Cardiac Arrest
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low enrollment
Sponsor: Jonathan Elmer (Other)
Collaborators: Laerdal Foundation (Other)
Responsible Party: Sponsor-Investigator, Jonathan Elmer, Assistant Professor, Department of Emergency Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO13060260
Record Dates: First submitted 2014-02-17; First posted 2014-02-24 (Estimated); Results first posted 2019-10-08 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-09

CONDITIONS: Cardiac Arrest
Keywords: Cardiac arrest; Neurological injury; Seizures; Spreading depolarizations; Cerebral hypoperfusion; Brain tissue hypoxia
MeSH Terms: conditions — Heart Arrest; Trauma, Nervous System; Seizures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cardiac arrest (Experimental): Survivors of cardiac arrest at high risk of neurological deterioration. Participants will undergo placement of a Spencer Probe Depth Electrode and QFlow 500™ Perfusion Probe in addition to the institutional standard multimodal neurological monitoring.
  Interventions: Device: QFlow 500™ Perfusion Probe (Hemedex, Cambridge, MA); Device: Spencer Probe Depth Electrode (Ad-Tech Medical, Racine, WI)

INTERVENTIONS:
Device: QFlow 500™ Perfusion Probe (Hemedex, Cambridge, MA)
Device: Spencer Probe Depth Electrode (Ad-Tech Medical, Racine, WI)

SUMMARY:
Cardiac arrest is the most common cause of death in the United States and as many as 590,000 Americans suffering a cardiac arrest each year. Despite advances in care, as many as 50 to 89% of patients who are resuscitated after a cardiac arrest die in the hospital. Brain injury is the most common cause of death and disability after cardiac arrest. The investigators use advanced brain monitoring in patients who are at high risk of death after cardiac arrest, with the goal of preventing ongoing brain injury. The most common problem the investigators have observed is low oxygen levels in the brain, which is often very difficult to treat.

In this study, the investigators plan to use two additional brain monitors in the care of these high risk patients: a monitor for seizures and a monitor of the amount of blood flow in the brain. The investigators will use these to detect and treat potential causes of low brain oxygen levels. The main hypotheses are that electrical events in the brain such as seizures and "spreading depolarizations" will occur during times of low brain tissue oxygen level, and that treating these events and low blood flow will reduce the rate of low brain oxygen levels.

ELIGIBILITY:
Inclusion Criteria:

* High risk survivors of cardiac arrest
* Decision by potential subject's clinical team to use our institutional standard invasive, multimodal neurologic monitoring for post-arrest care

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2015-07; Primary Completion 2018-10-19 (Actual); Study Completion 2018-10-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Cardiac Arrest: Survivors of cardiac arrest at high risk of neurological deterioration. Participants will undergo placement of a Spencer Probe Depth Electrode and QFlow 500™ Perfusion Probe in addition to the institutional standard multimodal neurological monitoring.
  QFlow 500™ Perfusion Probe (Hemedex, Cambridge, MA)
  Spencer Probe Depth Electrode (Ad-Tech Medical, Racine, WI)
Period: Overall Study
Arm/Group | Cardiac Arrest
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cardiac Arrest
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Spreading Depolarizations
Time Frame: Participants will be followed for the duration of invasive monitoring, an expected average of 5 days
Measure: Count of Participants; unit: Participants
Arm/Group | Cardiac Arrest
Number analyzed (Participants) | 4
Participants | 0

2. Primary Outcome: Occult Seizures
Description: Seizures detected by intracortical EEG but not surface EEG
Time Frame: Participants will be followed for the duration of invasive monitoring, an expected average of 5 days
Measure: Count of Participants; unit: Participants
Arm/Group | Cardiac Arrest
Number analyzed (Participants) | 4
Participants | 0

3. Primary Outcome: Cerebral Hypoperfusion
Time Frame: Participants will be followed for the duration of invasive monitoring, an expected average of 5 days
Measure: Count of Participants; unit: Participants
Arm/Group | Cardiac Arrest
Number analyzed (Participants) | 4
Participants | 4

4. Secondary Outcome: Clinically Significant Bleeding
Time Frame: Participants will be followed for the duration of the initial hospitalization, an expected average of 2 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Cardiac Arrest
Number analyzed (Participants) | 4
Participants | 0

5. Secondary Outcome: Monitor-associated Infection
Time Frame: Participants will be followed for the duration of the initial hospitalization, an expected average of 2 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Cardiac Arrest
Number analyzed (Participants) | 4
Participants | 0

6. Secondary Outcome: Device Malfunction
Time Frame: Participants will be followed for the duration of invasive monitoring, an expected average of 5 days
Measure: Count of Participants; unit: Participants
Arm/Group | Cardiac Arrest
Number analyzed (Participants) | 4
Participants | 0

ADVERSE EVENTS:
Time Frame: Duration of index hospitalization, a median of 3 days.
Description: Patients were examined by a study investigator daily to assess for adverse events until death or discharge.
Arm/Group | Cardiac Arrest
All-Cause Mortality (participants affected / at risk) | 3/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-30): https://cdn.clinicaltrials.gov/large-docs/53/NCT02069353/Prot_SAP_000.pdf